CLINICAL TRIAL: NCT06556511
Title: Khasiat Pemberian Zinc Terhadap Outcome Pada Anak Dengan Sepsis
Brief Title: Efficacy Of Zinc Towards The Outcome on Children With Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: dr. Aldora Jesslyn Oentari (Other)
Collaborators: Hasanuddin University (Other)
Responsible Party: Sponsor-Investigator, dr. Aldora Jesslyn Oentari, resident doctor, Hasanuddin University
Organization: Hasanuddin University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Zinc and Placebo
Record Dates: First submitted 2024-07-23; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Sepsis
Keywords: Sepsis; Zinc
MeSH Terms: conditions — Sepsis | interventions — Zinc Sulfate

STUDY DESIGN:
Intervention Model Description: Children with diagnosis of sepsis age 1 month to 18 years. Patients were divided into two groups, namely zinc group which received standard therapy with zinc, and placebo group which received standard therapy with placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- zinc group (Experimental): Children with diagnosis of sepsis. Patients who received standard therapy with zinc for 10 days
  Interventions: Drug: Zinc Sulfate
- placebo group (Placebo Comparator): Children with diagnosis of sepsis. Patients who received standard therapy with placebo for 10 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zinc Sulfate — Zinc is administered at a dose of 10 mg per day for children under the age of 6 months, and 20 mg per day for children above the age of 6 months accompanied with standard therapy in the zinc group for a period of 10 days.
  Other Names: zinc group
  Arms: zinc group
Drug: Placebo — Placebo is administered with standard therapy in the placebo group for a period of 10 days.
  Other Names: placebo group
  Arms: placebo group

SUMMARY:
Sepsis is a life-threatening organ failure induced by a compromised immune response to infection. Sepsis is a leading cause of morbidity and mortality (50-60%) in children treated in inpatient and critical care units. Children suffering from immunodeficiency have a higher mortality rate. Several studies in recent years have revealed that zinc homeostasis may be a significant role in the prevention of sepsis. It was important to conduct this study to determine the efficacy of zinc in children suffering from sepsis.

DETAILED DESCRIPTION:
This research is a randomized controlled trial with parallel study design conducted in Makassar, South of Sulawesi, Indonesia from February to May 2024. This study was conducted on children with a diagnosis of sepsis. Patients were divided into two groups, namely zinc group which received standard therapy with zinc and placebo group which received standard therapy with placebo.

The inclusion criteria were children aged 1 month to 18 years, diagnosed with sepsis, and parents/caregivers willing to participate their children in this study. Patients with diarrhea, malnutrition, Acute Kidney Injury due to kidney illness, hematological diseases, patients who have received zinc in the previous month, and patients who leave on their own request are all excluded from this study. Patients who not taking medication for up to three days in a row, either due to forgetfulness or self-determination, or due to side effects, and being unable to complete the study before the end date for various reasons, including death were declared dropouts.

Researchers will provide informed consent to parents/caregivers of children who met the research criteria. Anamnesis, general physical examination, and clinical also laboratory parameters were examined on day 0, 8, and 11 after zinc and placebo supplementation, such as; degree of consciousness, use of mechanical ventilators, P/F ratio, MAP, lactate levels, serum leukocyte and platelet counts, CRP and procalcitonin levels, lactate levels, sepsis progression, and mortality rates. The research results are recorded in a research form and the data is grouped and SPSS version 21.0 software is used for data analysis. A p value <0.05 was considered for statistical analysis. This study was approved by the ethics and research committee of the faculty of medicine, at Hasanuddin University.

ELIGIBILITY:
Inclusion Criteria:

- Children aged 1 month to 18 years with diagnosis of sepsis

Exclusion Criteria:

* Diarrhea
* Malnutrition
* Acute Kidney Injury due to kidney illness
* Hematological diseases
* Have received zinc in the previous month
* Leave on their own request

Dropping out criteria:

* Not taking medication for up to three days in a row
* Death

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
This study was to compare the effectiveness of standard therapy with zinc in children with sepsis | 10 days
  Comparing the level of awareness, used of a mechanical ventilator, P/F ratio, Mean Arterial Pressure (MAP), serum leukocytes and platelets, C-Reactive Protein (CRP) and procalcitonin levels, lactate levels, sepsis progression, and patient mortality between zinc group and placebo group on day 0, 8, and 11

SECONDARY OUTCOMES:
Comparing the mean changes in clinical and laboratory parameters | 10 days
  1. Comparing the difference of level of awareness, used of a mechanical ventilator, P/F ratio, Mean Arterial Pressure (MAP), serum leukocytes and platelets, C-Reactive Protein (CRP) and procalcitonin levels, lactate levels, sepsis progression, and patient mortality after treatment between zinc group and placebo group
  2. Comparing the difference of level of awareness, used of a mechanical ventilator, P/F ratio, Mean Arterial Pressure (MAP), serum leukocytes and platelets, C-Reactive Protein (CRP) and procalcitonin levels, lactate levels, sepsis progression, and patient mortality before and after treatment in the zinc group
  3. Comparing the difference of level of awareness, used of a mechanical ventilator, P/F ratio, Mean Arterial Pressure (MAP), serum leukocytes and platelets, C-Reactive Protein (CRP) and procalcitonin levels, lactate levels, sepsis progression, and patient mortality before and after treatment in the zinc group

CONTACTS AND LOCATIONS:
Overall Officials: Aldora Jesslyn Oentari, Principal Investigator — Hasanuddin University
Locations (1):
- Hasanuddin University, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No